CLINICAL TRIAL: NCT06528249
Title: Safety, Tolerability and Preliminary Efficacy of Erythrocyte-αPD-1 Conjugate Injection in Patients With Advanced Malignancies
Brief Title: Safety, Tolerability and Preliminary Efficacy of Erythrocyte-αPD-1 Conjugate in Patients With Advanced Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Westlake Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WTX212-002CN
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Solid Tumor; Hematologic Malignancy
Keywords: Cancer; Solid Tumor; Hematologic Malignancy
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, open-label, multicenter, multidose, dose escalation and expansion study to evaluate the safety, tolerability, and efficacy of Erythrocyte-αPD-1 conjugates in patients with advanced malignancies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Dose Escalation of Erythrocyte-αPD-1 conjugate monotherapy in patients with advanced malignancy
  Interventions: Drug: Engineered erythrocytes (or red blood cells) covalently conjugated with commercially available anti-PD-1 antibodies on their membranes
- Dose Expansion (Experimental): Dose Expansion of Erythrocyte-αPD-1 conjugate monotherapy in patients with advanced malignancy
  Interventions: Drug: Engineered erythrocytes (or red blood cells) covalently conjugated with commercially available anti-PD-1 antibodies on their membranes

INTERVENTIONS:
Drug: Engineered erythrocytes (or red blood cells) covalently conjugated with commercially available anti-PD-1 antibodies on their membranes — Engineered erythrocytes (or red blood cells) covalently conjugated with commercially available anti-PD-1 antibodies on their membranes

SUMMARY:
This is an investigator-initiated, multi-center, open-label clinical study to evaluate the safety, pharmacokinetics, pharmacodynamics, and efficacy of Erythrocyte-αPD-1 conjugates in patients with advanced malignancies

DETAILED DESCRIPTION:
This is an investigator-initiated, multi-center, open-label clinical study to evaluate the safety, pharmacokinetics, pharmacodynamics, and efficacy of Erythrocyte-αPD-1 conjugates in patients with unresectable or metastatic advanced malignancies who have failed previous systemic therapy.

The study was divided into two phases: dose escalation and dose expansion

ELIGIBILITY:
Inclusion Criteria:

1. The subject signs an informed consent form, understands this study, is willing to follow and has the ability to complete all experimental procedures;
2. Regardless of gender, aged 18 to 75 years old (including threshold);
3. Patients with advanced malignant tumors who have been confirmed by histopathology;
4. Patients with histopathologically confirmed unresectable or metastatic solid tumors who have failed systemic treatment or have no effective standard treatment, or who are unwilling to accept standard treatment or are not suitable for standard treatment;
5. ECOG≤1；
6. Expected life ≥ 3 months；
7. Male participants, their spouses, and female participants of childbearing age should agree to use a medically recognized effective contraceptive method from the signing of the informed consent form until 3 months after the last administration; Pregnancy testing results for women of childbearing age within ≤ 7 days before the first trial drug administration must be negative. Women of childbearing age include premenopausal women and women within 2 years after menopause.

Exclusion Criteria:

1. People with other serious medical diseases, including but not limited to: uncontrolled diabetes, active peptic ulcer, active bleeding, etc., and people with uncontrollable or serious cardiovascular diseases,
2. Patients with clinical symptoms and the need for repeated drainage of pleural and ascitic fluids;
3. Previous or recent history of pulmonary fibrosis, severe lung function damage caused by pneumoconiosis, radiation pneumonia, and drug-related pneumonia;
4. There have been adverse events related to the use of IO drugs that require permanent cessation of IO treatment;
5. Known to have other malignant tumors, currently progressing or completing treatment at least once in the past 3 years.
6. Subjects with symptomatic central nervous system (CNS) metastasis confirmed by imaging or pathological examination and clinically unstable for at least 14 days prior to enrollment who require steroid treatment;
7. Having hereditary bleeding tendencies or coagulation disorders, or a history of thrombosis, hemolysis, or hemorrhagic diseases; Received significant surgical treatment or obvious traumatic injury within 28 days prior to the start of research treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | through study completion, an average of 1 year
  The incidence of adverse events (AE), treatment related adverse events (TRAE), and severe adverse events (SAE) during the treatment of engineered erythrocytes

SECONDARY OUTCOMES:
Pharmacodynamics characteristics Peak Plasma Concentration(Cmax) | through study completion, an average of 1 year
  The occupancy rate of PD-1 receptor on the surface of peripheral blood T cells in subjects after infusion,including Peak Plasma Concentration(Cmax)
Pharmacodynamics characteristics Area under the plasma concentration versus time curve（AUC） | through study completion, an average of 1 year
  The occupancy rate of PD-1 receptor on the surface of peripheral blood T cells in subjects after infusion,including Area under the plasma concentration versus time curve (AUC).
Efficacy of Erythrocyte-αPD-1 Conjugate | per 6 weeks
  According to RECIST 1.1, the effectiveness of Erythrocyte-αPD-1 Conjugate injection in the treatment of patients with unresectable or metastatic advanced solid tumors was evaluated. The evaluation indicators included objective response rate (ORR),etc.

OTHER OUTCOMES:
Anti-drug antibody (ADA) | through study completion, an average of 1 year
  Describe the number of anti-drug antibodies (ADA) produced by subjects at each time point after treatment.
Peripheral immune response assessment | through study completion, an average of 1 year
  Immune cell alterations(number of T-cell,etc) in the peripheral are analyzed by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, PhD, Principal Investigator — ZHEJIANG PROVINCIAL PEOPLE'S HOSPITAL of China